CLINICAL TRIAL: NCT05876845
Title: A Clinical Trial to Assess the Effect of a Combined Pre-, Pro-, and Post-biotic Supplement on Gut and Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beekeeper's Naturals Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20291
Record Dates: First submitted 2023-04-20; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Gut Health
MeSH Terms: interventions — Proline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental)
  Interventions: Other: Combined pre-, pro-, and post-biotic supplement

INTERVENTIONS:
Other: Combined pre-, pro-, and post-biotic supplement — Participants will take 2 capsules daily with water, with their first meal of the day.

SUMMARY:
This is a virtual, single-arm clinical trial that will last 4-weeks. Participants will take the supplement daily and complete questionnaires at baseline, week 2, and week 4. Participants will provide photos of their face and stomach at baseline and week 4.

Gut health and associated health outcomes, including brain, skin, and immune function, will be evaluated at baseline and at each check-in. Likert scale responses will be statistically compared from baseline to each check-in. Participant responses on product feedback will be presented as % scores. Baseline and endline photos from each study part will be provided by participants.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* 18 years of age or older
* Experience at least one of the following symptoms: regular bloating/gas, irregular bowel movements, heartburn, or poor digestive health
* Generally healthy

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Allergic to bees, bee products, poplar tree products, or balsam of Peru
* Anyone with known severe allergic reactions.
* Women who are pregnant, breastfeeding or attempting to become pregnant
* Unwilling to follow the study protocol.
* Has introduced any new forms of medication or supplements targeting gut health within the last 3 months
* Has taken antibiotics in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Change in participant-reported gastrointestinal symptoms [Time Frame: Baseline to 4 weeks] | 4 weeks
  Assessed via study-specific questionnaires to gather information on improvements in bloating, digestion, stool regularity, stool quality, and gas. Survey-based assessments (0-5, 0-6 point scale) of changes in bloating, digestion, stool regularity, stool quality, and gas.
Change in scores on the Gastrointestinal Symptom Rating Scale (GSRS) [Time Frame: Baseline to 4 | 4 weeks
  Use of validated questionnaire the GSRS to assess gastrointestinal symptoms.The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters reporting on Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents no symptoms and 7 represents severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States